CLINICAL TRIAL: NCT05636826
Title: Efficacy of a Treatment Based on Olive Leaf Extracts in the Control of Cardiovascular Risk Factors:Hypertension
Brief Title: Olive Leaf Extracts in the Control of Hypertension
Acronym: Atherolive
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, clinical proffesor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATHEROLIVE-HTA
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Hypertension
Keywords: hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- atherolive-drug (Active Comparator): The patient will be assigned to one of two treatments (atherolive ) using a computer-generated randomization list (1: 1 allocation). The investigator who has the randomization code is not involved in other study procedures and does not interact with participants. The study drug (atherolive) will be prescribed at a dose of 400 mg, once a day for 3 months.
  Interventions: Drug: atherolive-drug
- atherolive-placebo (Placebo Comparator): The patient will be assigned to one of two treatments using a computer-generated randomization list (1: 1 allocation). The investigator who has the randomization code is not involved in other study procedures and does not interact with participants. The study drug (atherolive-placebo) will be prescribed at a dose of 400 mg, once a day for 3 months.
  Interventions: Drug: Placebo Atherolive

INTERVENTIONS:
Drug: atherolive-drug — The patient will be assigned to one of two treatments (atherolive ) using a computer-generated randomization list (1: 1 allocation). The investigator who has the randomization code is not involved in other study procedures and does not interact with participants. The study drug (atherol) will be prescribed at a dose of 400 mg, once a day for 3 months.
  Arms: atherolive-drug
Drug: Placebo Atherolive — The patient will be assigned to one of two treatments using a computer-generated randomization list (1: 1 allocation). The investigator who has the randomization code is not involved in other study procedures and does not interact with participants. Placebo will be prescribed at a dose of 400 mg, once a day for 3 months.
  Arms: atherolive-placebo

SUMMARY:
This study will be carried out in 2 emergency departments (at the exit of the emergency room) and 2 external consultations (endocrinology of the CHU FB Monastir and diabetology consultation, Jemmal hospital).

Patients over 18 years of age with:

Arterial hypertension (hypertension).

DETAILED DESCRIPTION:
This study will be carried out in 2 emergency departments (at the exit of the emergency room, patients included in the GR2 study) and 2 external consultations (endocrinology of the CHU FB Monastir and diabetology consultation, Jemmal hospital).

All the population will benifit of a biological assessment which include:

Complete lipid profile, blood sugar, creatinine

one population will be randomized:

The population of patients with hypertension.

For patients in the hypertension group:

A blood pressure with holter will be carried out for 24 hours .

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age with:

Arterial hypertension (hypertension)

Exclusion Criteria:

* . Exclusion criteria: None.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-12-30 (Actual); Primary Completion 2024-11-22 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
rate of blood pressure reduction | 90 days
  blood pressure reduction on 24 hours holter

SECONDARY OUTCOMES:
rate of lipid balance variation The secondary endpoint | 90 days
  variation in lipid reduction balance

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Fattouma Bourguiba Monastir, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No